CLINICAL TRIAL: NCT07126509
Title: A Pilot Study of Partial Pleurectomy in Borderline and Unresectable Pleural Mesothelioma
Brief Title: Partial Pleurectomy (Surgery) for Unresectable Pleural Mesothelioma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB25-1014
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Mesothelioma; Mesothelioma; Lung; Mesotheliomas Pleural; Mesothelioma Malignant Advanced; Mesothelioma, Malignant
Keywords: PLEURECTOMY
MeSH Terms: conditions — Mesothelioma; Mesothelioma, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All Study Participants (Experimental): This study arm will include all study participants receiving a partial pleurectomy (Surgery) for unresectable pleural mesothelioma. Participants in this study arm will all receive the same study procedures.
  Interventions: Procedure: Partial Pleurectomy

INTERVENTIONS:
Procedure: Partial Pleurectomy — A partial pleurectomy is a surgical procedure where part of the pleura, the lining of the lung cavity, is removed. This may be done to remove tumors, excess tissue, or to treat lung complications.

SUMMARY:
Purpose of the study: The main purpose of this research study is to see if a surgery procedure (limited partial pleurectomy and decortication) helps symptoms in people who have cancer that is unresectable that might not be able to be removed completely. This is called unresectable cancer. This study will also help the research team learn more about the types of symptoms and quality of life for people who have undergone this surgery, the number of complications following , and the time from surgery to starting other therapy. Th e study team also wants to see see the overall survival of people who have had this procedure as part of their care.

What will be done as part of research on this study:

* Surgery (Partial Pleurectomy - surgery to remove lining of lungs)
* The research team will also ask study participants questions about their symptoms through questionnaires at certain times after surgery.

How long this study will last:

Participation in this research (pre-surgery, surgery and follow-up) will last for about 2 years.

Confidentiality: All personal information will be kept confidential, and data will be used only for research purposes.

Contact Information: For more information about this study, please contact PhaseIICRA@medicine.bsd.uchicago.edu

ELIGIBILITY:
Inclusion Criteria

* Patients must have histologically confirmed epithelioid subtype pleural mesothelioma, as determined by surgical (i.e. VATS) biopsy.
* Disease confined to the unilateral hemithorax.
* Disease that is classified as unresectable or borderline resectable:
* Unresectable disease is defined by cross sectional imaging (CT or MRI) demonstrating invasion of unresectable mediastinal structures (heart, great vessels, esophagus) or spine, unresectable invasion of the chest wall (multifocal chest wall invasion or apical chest wall invasion), or disease outside intended resection field.
* Borderline resectable disease is defined by cross sectional imaging (CT or MRI) demonstrating extensive pulmonary parenchymal invasion (anticipated need for anatomic resection or complex wedge resection to clear disease) or extensive/bulky disease of (1) the diaphragm or sulci (anticipated need for diaphragm resection and reconstruction to clear disease), or (2) the chest wall (anticipated need for chest wall resection and reconstruction to clear disease). Disease with pathologically proven hilar or mediastinal lymph node involvement.
* Successful completion of at least 6 weeks of systemic induction therapy (regimen according to treating physician choice, including the below) with no unresolved adverse event that would preclude surgery:
* Platinum agent, pemetrexed, +/- bevacizumab
* Platinum agent, pemetrexed, pembrolizumab
* Ipilimumab/nivolumab
* Age ≥18 years.
* ECOG performance status ≤1.
* Patients must have adequate organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * PT/INR >1.5
  * PTT >Upper limit of normal
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification21. To be eligible for this trial, patients should be class 2B or better.
* Review by multidisciplinary treatment conference consisting of mesothelioma surgeons, radiologists, pathologists, medical oncologists, and palliative care physicians. Date of review will be documented in on the patient's elgibility checklist
* Prior or concurrent enrollment to UChicago's Mesothelioma Biobank (IRB15-0443).
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

* Patients with biphasic or sarcomatoid pleural mesothelioma.
* Patients with metastatic disease or disease which extends to the abdominal cavity or subdiaphragm as identified on post-induction therapy cross sectional imaging (CT, MRI, or PET).
* Patients who demonstrate disease progression during or following induction therapy.
* FEV1 < 50% and/or postoperative predicted DLCO < 50%.
* Patients who are receiving any other investigational agents.
* Patients with uncontrolled intercurrent illness.
* Prior malignancy active 2 years prior to registration except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast, or papillary thyroid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease-related Symptom Burden 3 Months After Partial Pleurectomy (Surgery) | 3 months after surgery
  The primary objective is to assess the post-operative disease-related symptom burden in participants undergoing partial pleurectomy and decortication for borderline or unresectable pleural mesothelioma, as measured by the mesothelioma-specific Lung Cancer Symptom Scale Average Symptom Burden Index (LCSS-meso ASBI) at 3 months post-surgery.

SECONDARY OUTCOMES:
Quality of Life of Study Participants Who Have Undergone Partial Pleurectomy (Surgery) | 2 years
  To longitudinally evaluate quality of life in patients who have undergone partial pleurectomy and decortication as assessed by quality of life questionnaires and patient reported outcomes.
Rate of Complications after Partial Pleurectomy (Surgery) | 2 years
  To estimate the rate of complications following partial pleurectomy and decortication as assessed by treating investigator and clinical notes.
Time to Resumption of Systemic Therapy | 2 years
  To determine time to resumption of systemic therapy following partial pleurectomy and decortication as assessed by treating investigator and clinical notes.
Overall Survival of Study Participants Who Have Undergone Partial Pleurectomy (Surgery) | 2 years
  To estimate overall survival in participants who have undergone partial pleurectomy and decortication as assessed by treating investigator and clinical notes.

CONTACTS AND LOCATIONS:
Overall Officials: Darren Bryan, MD, Principal Investigator — University of Chicago

IPD SHARING:
Plan to Share IPD: Undecided